CLINICAL TRIAL: NCT01825967
Title: Predictive Value of C-Reactive Protein in Acute Diverticulitis
Brief Title: Acute Diverticulitis and C-Reactive Protein as a Prognostic Marker
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, LAURA MORA LOPEZ, General Surgeon, Corporacion Parc Tauli
Other Study IDs: 2013/532
Record Dates: First submitted 2013-03-29; First posted 2013-04-08 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Acute Diverticulitis
MeSH Terms: interventions — C-Reactive Protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Diverticulitis: We measured C-reactive protein in all the patients diagnosed with acute diverticulitis
  Interventions: Other: C-reactive protein

INTERVENTIONS:
Other: C-reactive protein — measured C-reactive protein in all patients with acute diverticulitis

SUMMARY:
The management of acute diverticulitis maybe better if we have prognostic markers of evolution.

Hypothesis: C-reactive protein maybe a good prognostic marker of evolution of acute diverticulitis.

The investigators need to know the values of C-reactive protein to predict evolution of acute diverticulitis.

DETAILED DESCRIPTION:
A prospective observational study. All the patients with TC-diagnosis of acute diverticulitis (AD) had a C-reactive protein (PCR) in the initial blood test.

The investigators will predict evolution of AD with the PCR initial.

ELIGIBILITY:
Inclusion Criteria:

* Acute Diverticulitis

Exclusion Criteria:

* Other Abdominal Pathologies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients with Acute Diverticulitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: MORA LAURA, MD, Principal Investigator — Corporacion Parc Tauli
Locations (3):
- Spain (3):
  - Corporacion Parc Tauli, Sabadell, Barcelona
  - Corporacion parc tauli, Sabadell, Sabadell-Barcelona
  - Corporacion Parc Tauli, Sabadell, Sabadell/barcelona